CLINICAL TRIAL: NCT02619214
Title: Oxidative Stress Related to 2 Different Oxygen Concentrations During General Anesthesia. Clinical Trial.
Acronym: OSGA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-OXI-2013-62
Record Dates: First submitted 2015-11-25; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Oxidative Stress
Keywords: Oxidative Stress; Oxygen; General Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen 30% (Experimental): Patient receives 1 hour of general anesthesia with a 30% oxygen concentration.
  Interventions: Drug: 30% of oxygen concentration.
- Oxygen 60% (Experimental): Patient receives 1 hour of general anesthesia with a 60% oxygen concentration.
  Interventions: Drug: 60% of oxygen concentration.

INTERVENTIONS:
Drug: 30% of oxygen concentration. — 30% oxygen concentration during one hour of general anesthesia.
  Arms: Oxygen 30%
Drug: 60% of oxygen concentration. — 60% oxygen concentration during one hour of general anesthesia.
  Arms: Oxygen 60%

SUMMARY:
Clinical trial controlled randomized of parallels groups. The study is designed to look for differences in the oxidative stress level among healthy patients receiving 2 different oxygen concentrations: 30% and 60% during general anesthesia. Once the patient has been informed, the affirmative agreement has been obtained and inclusion and exclusion criteria verified the patients are randomized to 30% or 60% oxygen concentration. In the operating room while placing the intravenous line, a sample blood is obtained. General anesthesia is induced and maintained with sevoflurane. After Anesthesia induction the anesthesia machine is fixed in order to provide the oxygen concentration according to the randomization. One hour later a second venous sample is obtained. Samples are stored in cold conditions until their analysis in the laboratories of the biology faculty - Barcelona University.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery, under general anesthesia.
* ASA 1 - 2
* Orl surgery, reconstructive surgery, neck surgery, abdominal wall surgery.

Exclusion Criteria:

* Smoking Habit
* Pregnancy
* No compensated disease.
* ASA 3 or Higher.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in Malondialdehyde level | Baseline and after one hour of general anesthesia
  A blood sample is obtained before general anesthesia and a second sample is obtained one hour after the oxygen concentration has been fixed in the anesthesia machine.

SECONDARY OUTCOMES:
Change in proteic oxidation level | Baseline and after one hour of general anesthesia.
  A blood sample is obtained before general anesthesia and a second sample is obtained one hour after the oxygen concentration has been fixed in the anesthesia machine.
Change in glutathion level | Baseline and after one hour of general anesthesia.
  A blood sample is obtained before general anesthesia and a second sample is obtained one hour after the oxygen concentration has been fixed in the anesthesia machine.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Castrillon, M.D., Principal Investigator — Anesthesiologist.
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

REFERENCES:
- [Result] Finkel T, Holbrook NJ. Oxidants, oxidative stress and the biology of ageing. Nature. 2000 Nov 9;408(6809):239-47. doi: 10.1038/35041687. PMID 11089981
- [Result] Phillips M, Cataneo RN, Greenberg J, Grodman R, Gunawardena R, Naidu A. Effect of oxygen on breath markers of oxidative stress. Eur Respir J. 2003 Jan;21(1):48-51. doi: 10.1183/09031936.02.00053402. PMID 12570108
- [Result] Loiseaux-Meunier MN, Bedu M, Gentou C, Pepin D, Coudert J, Caillaud D. Oxygen toxicity: simultaneous measure of pentane and malondialdehyde in humans exposed to hyperoxia. Biomed Pharmacother. 2001 Apr;55(3):163-9. doi: 10.1016/s0753-3322(01)00042-7. PMID 11325214
- [Result] Winter PM, Smith G. The toxicity of oxygen. Anesthesiology. 1972 Aug;37(2):210-41. doi: 10.1097/00000542-197208000-00010. No abstract available. PMID 4559456
- [Result] Morita S, Snider MT, Inada Y. Increased N-pentane excretion in humans: a consequence of pulmonary oxygen exposure. Anesthesiology. 1986 Jun;64(6):730-3. doi: 10.1097/00000542-198606000-00009. PMID 3717636
- [Result] Griendling KK, FitzGerald GA. Oxidative stress and cardiovascular injury: Part I: basic mechanisms and in vivo monitoring of ROS. Circulation. 2003 Oct 21;108(16):1912-6. doi: 10.1161/01.CIR.0000093660.86242.BB. No abstract available. PMID 14568884
- [Result] Galley HF. Oxidative stress and mitochondrial dysfunction in sepsis. Br J Anaesth. 2011 Jul;107(1):57-64. doi: 10.1093/bja/aer093. Epub 2011 May 19. PMID 21596843
- [Result] Alonso de Vega JM, Diaz J, Serrano E, Carbonell LF. Plasma redox status relates to severity in critically ill patients. Crit Care Med. 2000 Jun;28(6):1812-4. doi: 10.1097/00003246-200006000-00021. PMID 10890625
- [Result] Alonso de Vega JM, Diaz J, Serrano E, Carbonell LF. Oxidative stress in critically ill patients with systemic inflammatory response syndrome. Crit Care Med. 2002 Aug;30(8):1782-6. doi: 10.1097/00003246-200208000-00018. PMID 12163793
- [Result] Khaw KS, Wang CC, Ngan Kee WD, Pang CP, Rogers MS. Effects of high inspired oxygen fraction during elective caesarean section under spinal anaesthesia on maternal and fetal oxygenation and lipid peroxidation. Br J Anaesth. 2002 Jan;88(1):18-23. doi: 10.1093/bja/88.1.18. PMID 11883375
- [Result] Khaw KS, Ngan Kee WD, Chu CY, Ng FF, Tam WH, Critchley LA, Rogers MS, Wang CC. Effects of different inspired oxygen fractions on lipid peroxidation during general anaesthesia for elective Caesarean section. Br J Anaesth. 2010 Sep;105(3):355-60. doi: 10.1093/bja/aeq154. Epub 2010 Jun 24. PMID 20576633
- [Result] Allaouchiche B, Debon R, Goudable J, Chassard D, Duflo F. Oxidative stress status during exposure to propofol, sevoflurane and desflurane. Anesth Analg. 2001 Oct;93(4):981-5. doi: 10.1097/00000539-200110000-00036. PMID 11574369
- [Result] Yagi K. Lipid peroxides and human diseases. Chem Phys Lipids. 1987 Nov-Dec;45(2-4):337-51. doi: 10.1016/0009-3084(87)90071-5. PMID 3319232
- [Result] Witko-Sarsat V, Friedlander M, Capeillere-Blandin C, Nguyen-Khoa T, Nguyen AT, Zingraff J, Jungers P, Descamps-Latscha B. Advanced oxidation protein products as a novel marker of oxidative stress in uremia. Kidney Int. 1996 May;49(5):1304-13. doi: 10.1038/ki.1996.186. PMID 8731095